CLINICAL TRIAL: NCT06743815
Title: Predictors of AKI in Patient Undergoing Colonoscopy
Brief Title: The Percent of AKI Occurred in Patient with Comorbidities Undergoing Colonoscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abd Elbasset Abd Elmoula Ahmed, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: AKI and colonoscopy; aki and colonoscopy (Other: Assiut University)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injuries
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- group: patients subjective for colonoscopy

SUMMARY:
observation the percent AKI in patient with comorbidities undergoing colonoscopy

DETAILED DESCRIPTION:
recording the data of the patient if there are any comorbidities like DM or HTN and observation of the kidney functions before and after the colonoscopy to record the percent of the AKI in patient undergoing colonoscopy

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged >18 years old Patient with eGFR>30ml/min

Exclusion Criteria:

* patient with eGFR <30ml/min patient with serum electrolytes abnormalities patient with heart diseases (uncontrolled heart failure, unstable angina, myocardial infarction, coronary intervention within the previous 3 months) patients with ascites

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient >18 years old with eGFR.30ml/min
Sampling Method: Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
incidence of acute kidney injury | 30 day
  the incidence of acute kidney injury in patients undergoing colonoscopy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Florentin M, Liamis G, Elisaf MS. Colonoscopy preparation-induced disorders in renal function and electrolytes. World J Gastrointest Pharmacol Ther. 2014 May 6;5(2):50-4. doi: 10.4292/wjgpt.v5.i2.50. PMID 24868484